CLINICAL TRIAL: NCT05601128
Title: An Open-label Study Evaluating the Pharmacokinetics (PK), Efficacy, Safety, and Tolerability of CABENUVA (Long-acting Cabotegravir Plus Long-acting Rilpivirine) Intramuscular (IM) Administered Monthly and Every 2 Months in Virologically Suppressed HIV-1-Infected Adults With Severe Renal Impairment With or Without Hemodialysis (CAPRI)
Brief Title: A Study Evaluating the Pharmacokinetics, Efficacy, Safety and Tolerability of CABENUVA
Acronym: CAPRI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Chiu-Bin Hsiao, MD, Physician, Physician Investigator, Medical Director Positive Health Clinic, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPRI
Record Dates: First submitted 2022-06-21; First posted 2022-11-01 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: HIV-1-infection; HIV Infections; HIV I Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIV + severe renal impairment (Experimental): CAB LA + RPV LA administered to HIV virologically suppressed participants with CKD stage 4/5 (CrCl < 30 mL/min) with (n = 6) or without (n = 6) hemodialysis receiving CABENUVA monthly for 6 months followed by every 2 months for 6 months.
  Interventions: Drug: CAB + RPV

INTERVENTIONS:
Drug: CAB + RPV — At Day 1 all participants will initiate oral CAB 30 mg + RPV 25 mg once daily for at least 28 days during the Oral Phase. Participants will receive CAB LA 600 mg + RPV LA 900 mg IM injections at month 1 visit followed by CAB LA 400 mg + RPV LA 600 mg IM injections monthly at M2, M3, M4 and M5 visits. Then, starting at month 6 visit, participants will receive CAB LA 600 mg + RPV LA 900 mg IM injections every 2 months at M6, M8, M10 and M12.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of CABENUVA (Long-acting Cabotegravir Plus Long-acting Rilpivirine) in patients with HIV infection and severe renal impairment. This study is considered research and is voluntary.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate CABENUVA (Long-acting Cabotegravir (CAB) Plus Long-acting Rilpivirine (RPV)) pharmacokinetics (movement of drugs within the body), safety and control of HIV in participants with renal (kidney) disease compared to historical values observed in those with normal renal function. Giving these drugs as an injection in your muscle (intramuscular) may offer be better tolerated by the body and may be simpler than taking a regular oral medication.

Researchers want to find out if two drugs long-acting CABENUVA can help people with HIV and kidney disease when given every 8 weeks (2 months) or every 4 weeks (monthly). 12 patients will be enrolled into this study between two study sites.

For the purposes of this project, we have applied for and received an FDA IND exemption (IND #161158) as this is a pilot study and not intended to result in a change in product labeling.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, at the time of signing the informed consent.
2. A female participant is eligible to participate if she is not pregnant as confirmed by negative urine HCG test at screening and at each study visits), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as:

* Pre-menopausal females with one of the following:

  1. Documented tubal ligation
  2. Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion
  3. Hysterectomy
  4. Documented Bilateral Oophorectomy
* Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood test result of simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (see Appendix 6) from 30 days prior to the first dose of study medication, throughout the study, for at least 14 days after discontinuation of all oral study medications and for at least 52 weeks after discontinuation of CAB LA and RPV LA.

The investigator is responsible for ensuring that participants understand how to properly use these methods of contraception. The study-sanctioned contraceptive method should be used consistently, in accordance with the approved contraceptive product label, before dosing of study medication and during the study intervention period

For all participants receiving oral standard of care (SOC) treatment for HIV-1:

1. Must be on uninterrupted current regimen (either the initial or second ARV regimen) for at least 6 months prior to Screening.
2. Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: one within the 6 to 12-month window, and one within 6 months prior to Screening
3. Plasma HIV-1 RNA <50 c/mL at Screening

Exclusion Criteria:

1. Screening plasma HIV-1 RNA measurement > 50 c/mL
2. Within 6 months prior to Screening, any plasma HIV-1 RNA measurement > 200 c/mL
3. Women who are pregnant, breastfeeding or plan to become pregnant or breastfeed during the study
4. Participants with severe hepatic impairment (Class C) as determined by Child-Pugh classification
5. Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant
6. Participants who, in the investigator's judgment, pose a significant suicide risk as assessed via the Columbia Suicidality Severity Rating Scale (C-SSRS). In addition, participant's recent history of mental health, psychiatric history, suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
7. Evidence of active Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV DNA as follows:

   * Participants positive for HBsAg are excluded:
   * Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded, not excluded if HBV DNA is negative or not detected
   * Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded
8. Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; participants who are anticipated to require HCV treatment within 12 months must be excluded.
9. Participants with HCV co-infection will be allowed entry into this study if:

   1. Liver enzymes meet entry criteria
   2. HCV Disease has undergone appropriate work-up, and is not advanced, and will not require treatment prior to the Week 52 visit. Additional information (where available) on participants with HCV co-infection at screening should include results from any liver biopsy, fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment.
   3. In the event that recent biopsy or imaging data is not available or inconclusive, the Fib-4 score will be used to verify eligibility
   4. Fib-4 score >3.25 is exclusionary
   5. Fib-4 scores 1.45 - 3.25 will require review by site PI to ensure that participant does not have severe liver disease and severe renal dysfunction. Fibrosis 4 Score Formula: (Age x AST) / (Platelets x (sqr [ALT])
10. History of liver cirrhosis with or without hepatitis viral co-infection
11. Ongoing or clinically relevant pancreatitis
12. Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medications
13. History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during PK sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled
14. Current or anticipated need for chronic anti-coagulation or hereditary coagulation and platelet disorders such as hemophilia or Von Willebrand Disease. The exception are the use of low dose acetylsalicylic acid (≤325 mg) or if, clinically, is safe to hold the anticoagulant for 1-3 days prior to the target time of CABENUVA injections and to re-start it 12 hours after the IM injections (upon Pharmacist, cardiologist or hematologist opinion).
15. Any evidence of primary resistance based on the presence of any major known INI or NNRTI resistance-associated mutation, except for K103N, (IAS, 2015) by any historical resistance test result. Note: Prior genotypic resistance testing is not required but if available it must be documented to provide direct evidence of no preexisting exclusionary resistance mutations. Details regarding baseline or prior resistance data must be noted in the source documentation
16. Any verified Grade 4 laboratory abnormality except Creatinine level (See Appendix 11). A single repeat test is allowed during the Screening phase to verify a result
17. Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's participation in the study of an investigational compound
18. Alanine aminotransferase (ALT) >=5x ULN, OR ALT >=3xULN and bilirubin >=1.5xULN (with >35% direct bilirubin)
19. Exposure to an experimental drug or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study: Treatment with any of the following agents within 28 days of Screening:

    1. radiation therapy
    2. cytotoxic chemotherapeutic agents
    3. tuberculosis therapy with the exception of isoniazid (isonicotinylhydrazid, INH)
    4. Immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons. (Note: Participants using short-term (e.g., ≤21 days) systemic corticosteroid treatment; topical, inhaled, and intranasal corticosteroids are eligible for enrolment)
20. Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
21. Use of medications which are associated with Torsade de Pointes.
22. Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.
23. Unstable renal disease and/or anticipated need for renal transplant within 1 year of study entry.

Note: Any prohibited medications that decrease CAB or RPV concentrations should be discontinued for a minimum of four weeks or a minimum of three half-lives (whichever is longer) prior to the first dose and any other prohibited medications should be discontinued for a minimum of two weeks or a minimum of three half-lives (whichever is longer) prior to the first dose.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Cabotegravir plasma concentration over time | Month 2 through Month 12 (for Ctrough)
  Since this is primarily a pharmacokinetics study, this descriptive outcome will demonstrate plasma concentration measures (Ctrough) versus time profiles for CAB LA.
Cabotegravir plasma concentration over time | Month 2 through Month 12 (for Cmax)
  Since this is primarily a pharmacokinetics study, this descriptive outcome will demonstrate plasma concentration measures (Cmax) versus time profiles for CAB LA.
Cabotegravir area under the curve | Month 1through Month 2, Month 5 through Month 6, and Month 10 through Month 12 (for AUC)
  Since this is primarily a pharmacokinetics study, this descriptive outcome will demonstrate "Area Under the Curve (AUC)" calculations for CAB LA.
Rilpivirine plasma concentration over time | Month 2 through Month 12 (for Ctrough)
  Since this is primarily a pharmacokinetics study, this descriptive outcome will demonstrate plasma concentration measures (Ctrough) versus time profiles for RPV LA.
Rilpivirine plasma concentration over time | Month 2 through Month 12 (for Cmax)
  Since this is primarily a pharmacokinetics study, this descriptive outcome will demonstrate plasma concentration measures (Cmax) versus time profiles for RPV LA.
Rilpivirine area under the curve | Month 1through Month 2, Month 5 through Month 6, and Month 10 through Month 12 (for AUC)
  Since this is primarily a pharmacokinetics study, this descriptive outcome will demonstrate "Area Under the Curve (AUC)" calculations for RPV LA.
Cabotegravir plasma concentration comparison between patients with severe renal impairment and those without severe renal impairment | Month 2 through Month 12
  Analysis of CAB LA plasma concentration measures (Ctrough) from participants with severe renal impairment compared to those from historical participants without severe renal impairment.
Cabotegravir plasma concentration comparison between patients with severe renal impairment and those without severe renal impairment | Month 2 through Month 12
  Analysis of CAB LA plasma concentration measures (Cmax) from participants with severe renal impairment compared to those from historical participants without severe renal impairment.
Cabotegravir plasma concentration comparison between patients with severe renal impairment and those without severe renal impairment | Month 2 through Month 12
  Analysis of CAB LA plasma concentration measures (AUC) from participants with severe renal impairment compared to those from historical participants without severe renal impairment.
Rilpivirine plasma concentration comparison between patients with severe renal impairment and those without severe renal impairment | Month 2 through Month 12
  Analysis of RPV LA plasma concentration measures (Ctrough) from participants with severe renal impairment compared to those from historical participants without severe renal impairment.
Rilpivirine plasma concentration comparison between patients with severe renal impairment and those without severe renal impairment | Month 2 through Month 12
  Analysis of RPV LA plasma concentration measures (Cmax) from participants with severe renal impairment compared to those from historical participants without severe renal impairment.
Rilpivirine plasma concentration comparison between patients with severe renal impairment and those without severe renal impairment | Month 2 through Month 12
  Analysis of RPV LA plasma concentration measures (AUC) from participants with severe renal impairment compared to those from historical participants without severe renal impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Allegheny Health Network, Pittsburgh, Pennsylvania, United States